CLINICAL TRIAL: NCT05778370
Title: Correlation Between HBA1c Level and Thickness of Both Macula and Choroid in Patients With Type 2 Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Salma Gamal Nouby Mahmoud, Resident doctor at soad kafafi hospital, Assiut University
Other Study IDs: HBA1c and OCT Macula
Record Dates: First submitted 2023-03-04; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- Group 1: will include 15 patients (30 eyes) of age matched non-diabetic candidates (control group)
  Interventions: Device: Swept Source Optical Coherence Tomography(Topcon DRI Triton)
- Group 2: will include 15 patients (30 eyes) of diabetic patients with good glycemic control (HbA1c ≤7%),
  Interventions: Device: Swept Source Optical Coherence Tomography(Topcon DRI Triton)
- Group 3: will include 15 patients (30 eyes) of diabetic patients with poor glycemic control (HbA1c <7% (
  Interventions: Device: Swept Source Optical Coherence Tomography(Topcon DRI Triton)

INTERVENTIONS:
Device: Swept Source Optical Coherence Tomography(Topcon DRI Triton) — Topcon DRI Triton

SUMMARY:
Diabetic retinopathy (DR) is a frequent cause of visual impairment, and the leading cause of blindness in those of working age, but it develops silently along years, producing symptoms only in late stages.

DETAILED DESCRIPTION:
The risk of sight-threatening consequences can be reduced if the lesions are detected before irreversible damage to retinal function has developed .Patients with diabetes mellitus (DM) have many pathological changes in their macula as diabetic macular edema (DME), exudates, cysts, detachment and ischemia that cause impairment of vision.

DME is characterized by increased vascular permeability and deposition of hard exudates at the macula and can occur at any stage of DR. With the help of OCT, it is possible to quantify the macular thickness objectively and to follow the progression of DME quantitatively.

Currently, DME is classified as 'center involved' or 'non center involved' (referring to whether or not there is oedema i.e., CMT>250 μm at the fovea) based on OCT. Non-centre involved macular oedema is rarely symptomatic. However, as the oedema spreads to the central macula, patients usually experience progressive vision loss and treatment with anti-VEGF is recommended.

Also, DM can cause many pathological changes in the choroid as increased tortuosity, focal vascular dilatation, microaneurysms and nonperfused areas. Studies have analyzed choroidal thickness changes in DR using spectral domain optic coherence tomography. A number of studies have shown that choroidal thickness decreases as the diabetic retinopathy progresses.

Swept-source (SS) OCT is a variation of OCT that offers improvements in visualizing the vitreous, retina, and choroid at one image. The increased scan speeds, decreased signal attenuation, more comprehensive imaging, and deeper tissue penetration make SS-OCT ideal for capturing a wide range of views and studying structures below the retinal pigmented epithelium (RPE), especially the choroid.

Glycated haemoglobin (HbA1c) is measured primarily to identify the average plasma glucose concentration over prolonged periods and reflect the long-term control of hyperglycaemia. Higher levels of HbA1c increase the incidence of DME over a 10-year period in Wisconsin Epidemiology Study of Diabetic Retinopathy (WESDR). The Diabetes Control and Complication Trial (DCCT) and the UK Prospective Diabetic Study (UKPDS) both of which were randomized prospective studies showed that intensive glycaemic control and thus reduction of HbA1c levels are associated with a decrease in the rates of development and progression of DR and DME.

The use of HbA1c for the diagnosis of DM has been approved by the WHO based on a number of epidemiological studies showing that a threshold for increased prevalence of microvascular complications can be observed at HbA1c level of 6.5% .

Aim of the work To investigate the correlation between HbA1c levels in patients with type II diabetes mellitus on central macular thickness as well as central choroidal thickness using swept source optical coherence tomography.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with type II diabetes mellitus and their age above 30 years.

  * No history of any previous ocular surgery.

Exclusion Criteria:

1. Unregulated arterial blood pressure, or cardiovascular disorder.
2. Media opacity that affects posterior pole imaging by OCT
3. Hyperopia of 4 diopters (D)
4. Myopia of -6 D.
5. Age related macular degeneration and other retinal or choroidal pathologies.
6. Any history of previous eye surgery.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Patients with type II diabetes mellitus and their age above 30 years.
  2. healthy population above 30 (for control group)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-04-15 (Estimated); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between HBA1c level and thickness of both macula and choroid in patients with type II diabetes mellitus | baseline
  Taking oct record for diabetic patients already know their HBA1c level ( done within 3 months max ) . Without follow up Findings will be compared controlled and non controlled group and with control group (normal people) To correlate if there's relavence between the Hba1c and macular thickness

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S Saad, Prof, Study Chair — Assiut University; Mohamed Sharaf-Eldin, Dr, Study Director — Assiut University; Dalia M Ali, Dr, Principal Investigator — Assiut University